CLINICAL TRIAL: NCT06272136
Title: An Exploratory Study to Assess the Accuracy in the Normo- to Hyperglycemic Range of the Spiden Non-invasive Continuous Glucose Monitor "Clinical Demo" (niCGM), in Trial Participants with Type 1 or Type 2 Diabetes
Brief Title: Liom Non-invasive Continuous Glucose Monitor "Clinical Demo" (niCGM)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Liom Health AG (Industry)
Collaborators: Profil Institut für Stoffwechselforschung GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SPN-007
Record Dates: First submitted 2024-01-31; First posted 2024-02-22 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Type 1 Diabetes; Type2diabetes
Keywords: Hyperglycemia; Diabetes Mellitus; Transcutaneous; Spectral fingerprint; Non-invasive
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hyperglycemia; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Interventional arm (Experimental): Induction of hyperglycaemia and hypoglcemia states and measurements of transcutaneous spectral data with the investigational device and reference blood glucose values measured by Super GL and Freestyle Libre 3.
  Interventions: Device: Clinical Demo 2.0

INTERVENTIONS:
Device: Clinical Demo 2.0 — During the different glycaemia states, transcutaneous spectral data are collected continuously with the device and paired with reference measurements (venous blood and interstitial fluid)

SUMMARY:
This is a single-centre, multiple cohort, open study.

DETAILED DESCRIPTION:
The study will include 5 cohorts. After each cohort, optimisation of the Spiden Clinical Demo 2.0 system and machine learning models may be pursued before the next cohort is started. Trial participants with type 1 or type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Male or female trial participant with clinically diagnosed type 1 or type 2 diabetes for at least 1 year.
* Age between 18 and 65 years, both inclusive.
* Treated with insulin and/or oral antidiabetic drugs (OADs; type 2 only), multiple dosing insulin therapy (MDI), continuous subcutaneous insulin infusion (CSII) or a hybrid closed loop system.

Exclusion Criteria:

* Known or suspected hypersensitivity to any of the components of the Liom Clinical Demo 2.0.
* Trial participant with any injury, infection, atypical skin condition (e.g., hyperkeratosis, hyperpigmentation) of or tattoo on the wrists.
* Presence or history of a cardiovascular disease including stable and unstable angina pectoris, myocardial infarction, transient ischaemic attack, stroke, cardiac decompensation, clinically significant arrhythmias or clinically significant conduction disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-02-23 (Actual); Primary Completion 2025-07-21 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Glucose changes will be measured noninvasively and transcutaneously in dynamic states of glycaemia | The data is collected during the study procedure (up to 5 hours)
  Spectroscopic research platform and associated computational models will be used to detect and track glucose changes noninvasively and transcutaneously in dynamic states of glycaemia

CONTACTS AND LOCATIONS:
Overall Officials: Marc Stoffel, MD, Principal Investigator — Profil for Stoffwechselforschung GmbH, Neuss, Germany
Locations (1):
- Profil for Stoffwechselforschung GmbH, Neuss, Nordrhein-Westfallen, Germany

IPD SHARING:
Plan to Share IPD: No